CLINICAL TRIAL: NCT01270035
Title: Efficacy and Safety of Adalimumab 80 mg Every Other Week With Methotrexate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keio University (Other)
Collaborators: Saitama Medical University (Other)
Responsible Party: Hideto Kameda, Keio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADA80MTX
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

ARMS (1):
- ADA 80 mg eow + MTX (Experimental)
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — To increase the ADA dose from 40 mg eow to 80 mg eow

SUMMARY:
In Japan, as well as in other countries, the dose of adalimumab (ADA) is limited to 40 mg every other week when used in combination with methotrexate (MTX) for patients with rheumatoid arthritis (RA). However, ADA 80 mg with MTX may be required for some RA patients, especially for those with high disease activity. Therefore, we tried to increase the ADA dose to 80 mg every other week with concomitant MTX, only if the disease activity did not decrease below moderate activity defined by DAS28 < 3.2. The primary endpoint was the rate of patients who achieved disease remission (DAS28 < 2.6) at 30 weeks with this predifined treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* patients with rheumatoid arthritis receiving MTX ≧ 6 mg/week for at least 3 months disease activity : DAS28 > 5.1

Exclusion Criteria:

* allergy to ADA present active infection including TB history of demyelinating disease, HBV infection and malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
The rate of achieving remission at week 30 | 30 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Saitama Medical Center, Kawagoe, Saitama
  - Keio University Hospital, Shinanomachi, Tokyo